CLINICAL TRIAL: NCT07253883
Title: A Diagnostic Accuracy Study: N-Tidal Assessment for Respiratory Diagnosis Compared to Using Standard Testing
Brief Title: A Study to Understand the Accuracy of a New Breathing Device Compared to Standard Testing for Asthma and COPD
Acronym: STARDUST
Status: Not yet recruiting | Type: Observational
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: TidalSense (Industry)
Responsible Party: Sponsor
Other Study IDs: 1694
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Asthma (Diagnosis); COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Asthma; COPD; End tidal CO2; Diagnostics; Machine learning
MeSH Terms: conditions — Asthma; Disease; Pulmonary Disease, Chronic Obstructive | interventions — Fractional Exhaled Nitric Oxide Testing; Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Asthma: Patients with suspected asthma
  Interventions: Diagnostic Test: Partial pressure of CO2 during tidal breathing; Diagnostic Test: FENO; Diagnostic Test: Spirometry
- COPD: Patients with suspected COPD
  Interventions: Diagnostic Test: Partial pressure of CO2 during tidal breathing; Diagnostic Test: FENO; Diagnostic Test: Spirometry

INTERVENTIONS:
Diagnostic Test: Partial pressure of CO2 during tidal breathing — Partial pressure of CO2 during tidal breathing for diagnosis of asthma or COPD
Diagnostic Test: FENO — Fractional exhaled nitric oxide
  Other Names: Fractional exhaled nitric oxide
Diagnostic Test: Spirometry — Spirometry with or without bronchodilation (if indicated)

SUMMARY:
The diagnosis of either asthma or chronic obstructive pulmonary disease (COPD) is currently based on a combination of symptoms, different lung tests and sometimes a 'trial by treatment'. Both COPD and Asthma tests currently include forced breathing using a test known as spirometry which can be difficult and uncomfortable for people to perform and needs expert interpretation. Asthma can require multiple tests in sequence which can make the process of diagnosis long and inconvenient for patients. In the UK, there have been challenges providing enough testing for COPD and asthma, in part because the tests are challenging to provide in the community to everyone who needs one.

The STARDUST study aims to test and develop new ways of diagnosing asthma and COPD that are quick, accurate and easy for patient and healthcare professionals to perform. People who have been referred for routine lung testing will breathe normally in and out into a handheld device called the N-Tidal Handset for 75 seconds. This device measures how the level of carbon dioxide (CO2) changes in the breath as people breath through it. The information gathered on the N-Tidal Handsets, called breath records or capnograms, will not be used to alter the diagnosis of any participants in the study.

After the capnograms have been collected, the research team will test 'algorithms' that have been developed using artificial intelligence, to see if they can accurately identify the correct diagnosis. Information collected in the study will also be used to make improvements in these algorithms.

If confirmed to be accurate, these algorithms could be used in clinical practice to help healthcare professionals make faster, more accessible and accurate diagnoses, especially in settings like GP clinics in the community where access to specialist tests may be limited.

DETAILED DESCRIPTION:
COPD is one of the leading causes of disability and in the top five causes of death worldwide. Early diagnosis and treatment are essential to slow the decline of lung function and improve quality of life.

The current standard for diagnosing COPD is spirometry; an effort-dependent test that requires supervised use, by a specifically trained medical professional, in a clinic-based environment. It is estimated that up to 2/3 of cases are undiagnosed suggesting that there is a significant care gap in the ability to accurately diagnose COPD.

Asthma is a chronic respiratory disease, characterised by airway inflammation and hyper-responsiveness. In 2019 affected an estimated 262 million people. Early diagnosis and treatment are important to reduce symptoms, exacerbations and mortality and to improve overall quality of life. The confirmation of reversible airflow obstruction using pre- and post-bronchodilator (BD) spirometry is needed to confirm a diagnosis in those suspected as having asthma without evidence of inflammation in the airways or blood.

Spirometry can be challenging for patients to perform, is time consuming and can be challenging to deliver at the scale required by the population.

TidalSense have been developing respiratory diagnostic devices that could offer simpler, safe, fast, reliable and precise tests to diagnose both COPD and asthma.

It is anticipated that successfully meeting the primary objectives of this study will result in data on the diagnostic accuracy of the COPD diagnostic models and could lead to the development and improvement of all diagnostic algorithms used in the study. This may contribute to a range of future clinical benefits:

* Accurate diagnosis of asthma and/or COPD
* Accurate detection of severe COPD in patients who are likely or highly likely to have COPD
* Improved ease of testing for asthma and/or COPD for patients and healthcare professionals
* Clearer differentiation between asthma and COPD in patients with overlapping symptoms

These benefits could enable quicker testing, improve patient experience (relaxed breathing instead of forced breathing), and improve patient access to testing compared to current diagnostic pathways and reduce misdiagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Referred for respiratory diagnostic testing with a clinical suspicion of asthma or COPD
* Participant is willing and able to provide informed consent

Exclusion Criteria:

* Referred for respiratory diagnostic testing for a condition other than asthma or COPD, with no mention in the referral of a clinical suspicion of COPD or asthma
* Participants who, in the opinion of the chief investigator, or their delegate, are unlikely to comply with the requirements of the study
* Inability to give written informed consent
* Participants who are acutely unwell
* Patients unable to breathe through their mouths e.g. tracheostomy patients

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a suspicion of asthma and/or COPD
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-12-19 (Estimated); Study Completion 2027-05-19 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the diagnostic algorithms of N-Tidal Diagnose 1 | At time of testing
  PPV, NPV, Sensitivity, Specificity compared to clinician diagnosis of COPD
Diagnostic accuracy of prototype diagnostic algorithms | At time of testing
  Prototype asthma diagnostic algorithms (index test; PPV, NPV, Sensitivity, Specificity) trained using a combined capnogram dataset from this and previous studies, compared to clinician diagnosis of asthma

SECONDARY OUTCOMES:
Diagnostic accuracy of the N-Tidal Diagnose 1 severity algorithm | At time of diagnsosis
  Diagnostic accuracy (PPV, NPV, Sensitivity, Specificity) of the N-Tidal Diagnose 1 severity algorithm in those with a confirmed diagnosis of COPD. Diagnostic accuracy (PPV, NPV, Sensitivity, Specificity) of the diagnostic algorithms embedded in NTidal Diagnose 1 v1.0 in relevant subgroups. Diagnostic accuracy (PPV, NPV, Sensitivity, Specificity) of the pre-production asthma diagnostic algorithms trained using a combined capnogram dataset from this and previous studies in relevant prespecified subgroups. Exploratory analysis of novel machine learning diagnostic algorithms for COPD and asthma.
Feasibility and acceptability outcomes | At time of diagnosis
  Visual Analogue Score (VAS) following N-Tidal, spirometry and FeNO (ease of use and comfort for participants, ease of use only for administering healthcare professionals) in a subset of participants. Percentage of participants with a clinical suspicion of COPD with adequate N-Tidal Handset breath record capture, sufficient to generate a diagnostic output using N-Tidal Diagnose 1 v1.0 diagnostic algorithms. Percentage of participants with a clinical suspicion of asthma with adequate N-Tidal Handset breath record capture, sufficient to generate a diagnostic output using prototype asthma diagnostic algorithms.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared for future research under appropriate governance as per the terms of the collaboration agreement between TidalSense and the Liverpool Heart and Chest Hospital NHS Foundation Trust.